CLINICAL TRIAL: NCT00133887
Title: Efficacy of Rapamycin in Secondary Prevention of Skin Cancers in Kidney Transplant Recipients - Multicentric Randomized, Open-label Study of Rapamycin vs Calcineurin Inhibitors
Brief Title: TUMORAPA 1: Efficacy of Rapamycin in Secondary Prevention of Skin Cancers in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003.333
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Skin Cancer; Kidney Transplantation
Keywords: Squamous cell carcinoma; kidney transplant recipients; rapamycin; Skin cancers in kidney transplant recipients
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell | interventions — Sirolimus; Cyclosporins; Tacrolimus

ARMS (2):
- 1 (Experimental): patients receiving Rapamycin
  Interventions: Drug: rapamycin
- 2 (Active Comparator): patients receiving anticalcineurin treatment
  Interventions: Drug: ciclosporine; Drug: tacrolimus

INTERVENTIONS:
Drug: rapamycin — 3 to 5 mg/day
  Other Names: Rapamune
  Arms: 1
Drug: ciclosporine — Blood residual level < or = to 125 ng/ml
  Arms: 2
Drug: tacrolimus — Blood residual level < or = to 8 ng/ml
  Arms: 2

SUMMARY:
In a population of kidney transplant recipients having developed a first squamous cell carcinoma, the aim of the study is to assess the incidence of subsequent skin cancers over 2 years in patients who are switched to rapamycin as compared to patients who are maintained under calcineurin inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* First post-transplant squamous cell carcinoma in a kidney transplant recipient under calcineurin inhibitors

Exclusion Criteria:

* Other squamous cell carcinomas in the past history
* More than 2 transplantations
* Patients not under calcineurin inhibitors
* Unstable graft function
* Non controlled hyperlipidemia (cholesterol > 7.8 mmol/l or triglycerides > 3.95 mmol/l)
* Leucopenia < 3000/mm3
* Thrombocytopenia < 100,000/mm3
* Liver dysfunction
* Pregnancy
* Allergy to macrolides

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-04; Primary Completion 2011-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of new squamous cell carcinoma in kidney transplant recipients | during 5 years

SECONDARY OUTCOMES:
To assess the incidence of other non skin cancer in kidney transplant recipients | during 5 years
To assess the graft survival | during 5 years
To assess the tolerance of rapamycin | during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie EUVRARD, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - Service de Dermatologie, Lyon, France

REFERENCES:
- [Result] Dantal J, Morelon E, Rostaing L, Goffin E, Brocard A, Tromme I, Broeders N, Del Marmol V, Chatelet V, Dompmartin A, Kessler M, Serra A, Hofbauer GFL, Kamar N, Pouteil-Noble C, Kanitakis J, Roux A, Decullier E, Euvrard S; TUMORAPA Study Group. Sirolimus for Secondary Prevention of Skin Cancer in Kidney Transplant Recipients: 5-Year Results. J Clin Oncol. 2018 Sep 1;36(25):2612-2620. doi: 10.1200/JCO.2017.76.6691. Epub 2018 Jul 17. PMID 30016177
- [Result] Euvrard S, Morelon E, Rostaing L, Goffin E, Brocard A, Tromme I, Broeders N, del Marmol V, Chatelet V, Dompmartin A, Kessler M, Serra AL, Hofbauer GF, Pouteil-Noble C, Campistol JM, Kanitakis J, Roux AS, Decullier E, Dantal J; TUMORAPA Study Group. Sirolimus and secondary skin-cancer prevention in kidney transplantation. N Engl J Med. 2012 Jul 26;367(4):329-39. doi: 10.1056/NEJMoa1204166. PMID 22830463
- [Result] Aractingi S, Kanitakis J, Euvrard S, Le Danff C, Peguillet I, Khosrotehrani K, Lantz O, Carosella ED. Skin carcinoma arising from donor cells in a kidney transplant recipient. Cancer Res. 2005 Mar 1;65(5):1755-60. doi: 10.1158/0008-5472.CAN-04-2783. PMID 15753371
- [Result] Martinez JC, Otley CC, Euvrard S, Arpey CJ, Stasko T; International Transplant-Skin Cancer Collaborative. Complications of systemic retinoid therapy in organ transplant recipients with squamous cell carcinoma. Dermatol Surg. 2004 Apr;30(4 Pt 2):662-6. doi: 10.1111/j.1524-4725.2004.30153.x. PMID 15061852